CLINICAL TRIAL: NCT00086216
Title: An Open-Label Study of the Safety and Efficacy of Atiprimod Treatment for Patients With Refractory or Relapsed Multiple Myeloma
Brief Title: Safety and Efficacy of Atiprimod for Patients With Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Callisto Pharmaceuticals (Industry)
Responsible Party: Gary Jacob, Callisto Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-101; efficacy; pharmacokinetics; research markers; NCT00301977 (obsolete NCT alias); NCT00491972 (obsolete NCT alias)
Record Dates: First submitted 2004-06-28; First posted 2004-06-30 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — azaspirane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Atiprimod — Oral, once a day, 14 days on 14 days off

SUMMARY:
This is a Phase I/IIa clinical trial to identify the maximum tolerated dose of atiprimod and to evaluate the safety of atiprimod in patients with refractory or relapsed multiple myeloma.

DETAILED DESCRIPTION:
This is a multi-center, open-label, dose escalation study intended to identify the MTD of atiprimod alone and the MTD of atiprimod when given in combination with ursodiol. The atiprimod dose will be escalated in sequential cohorts. Ten dose levels of atiprimod are planned for the atiprimod alone dose escalation: 30, 60, 90, 120, 180, 240, 300, 360, 420, and 480 mg/day to be given orally. Six dose levels of atiprimod are planned for the atiprimod in combination with ursodiol dose escalation: 180, 240, 300, 360, 420, and 480 mg/day to be given orally. The dose of ursodiol will remain constant for all cohorts (300 mg ursodiol orally three times a day everyday). Up to 105 patients will participate depending on the level at which toxicity is observed. Patients will be assigned to dose level in the order of study entry.

ELIGIBILITY:
Inclusion Criteria:

* documented history of multiple myeloma,
* failed at least two prior regimens for multiple myeloma,
* 18 years of age or older,
* ECOG(Zubrod)PS of 0 to 2,
* screening evaluation for determining eligibility prior to enrollment,
* signed informed consent form,

Exclusion Criteria:

* concomitant therapy medications including corticosteroids or other chemotherapy that is or may be active against myeloma ,
* renal insufficiency (serum creatinine levels of > 2mg/dL),
* mucosal bleeding,
* any condition which in the opinion of the Investigator, places the patient at unacceptable risk if he/she were to participate in the study.
* clinically relevant active infection or co-morbid medical conditions.
* prior malignancy(within the last 3 years) except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient is has been disease-free for at least 3 years.
* patients with non-secretory myeloma.
* as atiprimod is a potent inhibitor or CYP2D6, patients taking drugs that are substrates of CYP2D6(e.g. beta blockers, antidepressants and antipsychotics) will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-05; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to identify the maximum tolerated dose | 1 year

SECONDARY OUTCOMES:
The secondary objective of this study is to measure the pharmacokinetics of | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gary Jacob, PhD, Study Director — Callisto Pharmaceuticals
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States